CLINICAL TRIAL: NCT06847191
Title: A Double-blind, Randomized Study to Evaluate the Efficacy and Safety of Bezisterim (NE3107) in Adults With Long COVID
Brief Title: NE3107 in Adults With Neurological Symptoms of Long COVID
Acronym: ADDRESS-LC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioVie Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NE3107-LC-201; CDMRP-PR230631 (Other Grant/Funding Number: DOD)
Record Dates: First submitted 2025-02-24; First posted 2025-02-26 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Long COVID
Keywords: COVID-19; Neurocognition; Fatigue; Post-exertional malaise; Sleep; SARS-CoV-2; Brain fog
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19; Fatigue; Mental Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant, investigator, assessors, or any member of the study staff at the CRO or sponsor will be masked to the treatment assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NE3107 (Experimental): One 20 mg capsule containing NE3107 taken by mouth twice daily (BID)
  Interventions: Drug: NE3107
- Placebo (Placebo Comparator): One 20 mg capsule containing placebo taken by mouth twice daily (BID)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NE3107 — 20 mg Capsule
  Other Names: bezisterim
  Arms: NE3107
Drug: Placebo — placebo capsule
  Arms: Placebo

SUMMARY:
Long COVID is a condition where debilitating symptoms can persist for months after a COVID-19 infection. This study aims to evaluate the effects of NE3107 on several neurological symptoms reported in people with Long COVID including difficulty concentrating or remembering things ("brain fog") and fatigue.

Researchers will compare NE3107 to a placebo (a look-alike substance that contains no drug) to see if NE3107 works to treat neurocognitive and fatigue symptoms of long COVID.

Participants will:

* Take NE3107 or a placebo twice daily for 84 days
* Visit the clinic 5 times for checkups and tests and have a follow up phone call

ELIGIBILITY:
Key Inclusion Criteria:

* 18 years to 69 years of age
* Long COVID with neurological symptoms as defined below:

  1. Current symptoms of at least fatigue and neurocognitive impairment that began or worsened after an index SARS-CoV-2 infection that occurred at least 3 months prior to screening. Index SARS-CoV-2 infection is defined as either: 1) an episode of COVID-19 with a positive nucleic acid or antigen test during acute illness, as documented in the medical record, or 2) a documented clinical diagnosis of COVID-19, which can be based on a patient-reported positive test for COVID-19. Note that a documented diagnosis of Long COVID is not required for inclusion.
  2. Symptoms cannot be explained by any concomitant condition or diagnosis, in the opinion of the investigator.
  3. Symptom duration for at least 3 months. diagnosed with Long COVID with symptoms of fatigue and brain fog for at least 3 months
* Agree to maintain any other regular medications at current doses for the duration of the trial (except for essential need of new medication or dose change, as prescribed by a physician)
* Agree to use birth control measures
* Provide voluntary consent
* Willing to allow blood collection
* Pass all screening tests and procedures

Key Exclusion Criteria:

* Has received a COVID-19 vaccination within 14 days
* Previous admission to the intensive care unit for COVID-19
* Medical history of major mental or physical illness prior to COVID-19 infection

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in performance on the Cogstate Cognition battery | 12 Weeks

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Stanford University, Palo Alto, California
  - UCSF, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Clinical Trial Site, Jacksonville, Florida
  - Centricity Research, Columbus, Georgia
  - Illinois Research Network University of Illinois at Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Norton Infectious Disease Institute, Louisville, Kentucky
  - Jadestone Clinical Research, Silver Spring, Maryland
  - Clinical Trial Site, Farmington Hills, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Zenos Clinical Research, Dallas, Texas
  - University of Texas health Science Center at San Antonio, San Antonio, Texas
  - Swedish Center for Research and Innovation, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ADDRESSLC Study website — https://addresslongcovid.com